CLINICAL TRIAL: NCT04448470
Title: Comparison Between the Situational and the Time-of-day Recording of Daytime Sleepiness in Patients With the Assessment of a Sleep-related Respiratory Disorder
Brief Title: Daytime Sleepiness in Patients With the Assessment of a Sleep-related Respiratory Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator Dr. Stefanie Keymel, Heinrich-Heine University, Duesseldorf
Other Study IDs: 19-002
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Sleep-related Respiratory Disorder
Keywords: daytime sleepiness; respiratory disorder; sleep apnea
MeSH Terms: conditions — Disorders of Excessive Somnolence; Respiration Disorders; Sleep Apnea Syndromes | interventions — Surveys and Questionnaires; Immunologic Memory; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with a clinical suspicion of sleep apnea (n=150): patients with a clinical suspicion of sleep apnea
  Interventions: Other: Questionnaire for recording daytime sleepiness over the course of the day; Other: Anamnesis and physicial examination; Other: Questionnaire for quantifying daytime sleepiness; Diagnostic Test: Pulmonary function test; Diagnostic Test: Polygraphy
- healthy subjects (n=10): healthy subjects
  Interventions: Other: Questionnaire for recording daytime sleepiness over the course of the day; Other: Anamnesis and physicial examination; Other: Questionnaire for quantifying daytime sleepiness; Diagnostic Test: Pulmonary function test; Diagnostic Test: Polygraphy

INTERVENTIONS:
Other: Questionnaire for recording daytime sleepiness over the course of the day — Questionnaire for recording daytime sleepiness over the course of the day
Other: Anamnesis and physicial examination — Anamnesis and physical examination, e.g. medication, comorbidities, complaints
Other: Questionnaire for quantifying daytime sleepiness — the Epworth Sleepiness Scale (ESS) questionnaire and the STOP BANG Questionnaire
Diagnostic Test: Pulmonary function test — The measured values of spirometry/body plethysmography, CO diffusion and blood gas analysis are documented, if available.
Diagnostic Test: Polygraphy — Polygraphy is a non-invasive portable examination method that the patient uses in the home environment at night to measure possible sleep-related breathing disorders. Typically, the following measurement signals are recorded: nasal airflow, thoracic and abdominal breathing excursions, snoring and breathing sounds via a microphone, pulse, oxygen saturation and position. The evaluation results and the findings are checked by a physician. Essential parameters include the apnoea-hypopnoea index, the number of obstructive, central and mixed apnoea/hypopnoea, the number and duration of desaturation, snoring or the association with a certain position.

SUMMARY:
It is not yet known whether an analysis of daytime sleepiness over the course of the day can predict the diagnosis or severity of sleep apnea. The goal of the study is to examine whether a psychometric determination of daytime sleepiness can adequately and practicably record daytime sleepiness in patients with mainly sleep apnea in comparison to other standardized methods.

DETAILED DESCRIPTION:
Detailed Description: Sleep-related respiratory disorders are a common disease in the general population. Untreated sleep apnea is associated with an increased risk of accidents, an increased risk of perioperative complications and various cardiovascular diseases such as arterial hypertension, coronary heart disease or stroke. Sleep apnea is often undetected. As part of the diagnosis of sleep apnea, screening is usually carried out to assess the probability of pre-testing before a sleep medical examination by means of anamnesis, examination and recording of risk factors and comorbidities. Questionnaires play a decisive role here. The Epworth Sleepiness Scale (ESS) or the STOP BANG questionnaires are often used for this purpose. ESS asks about the probability of falling asleep in different situations. With STOP BANG, the points daytime tiredness, snoring, breathing stops and various risk factors such as age, sex, neck circumference, high blood pressure and overweight are asked. The quality of the questionnaire used to assess the risk of sleep apnea is of crucial importance, as it is usually the basis for the decision whether or not to perform further sleep medical diagnostics. To date, there is no established, easy-to-use method for measuring daytime sleepiness during the day. However, it can be assumed that the degree of daytime sleepiness can predict the presence of sleep apnea. In a proof-of-concept study, the psychometric determination of daytime sleepiness in a time series on one day in patients with mainly sleep apnea will be measured.

The following questions should be answered:

1. Does daytime sleepiness in patients with sleep apnea measured by a scale-based, psychometric time-series test show one or more characteristic patterns over the day?
2. Is there a relation between the degree of the scale based psychometric time series test for daytime sleepiness and the severity of sleep apnea?
3. Is the test quality of the scale based psychometric time series test for predicting sleep apnea better than the established Epworth Sleepiness Scale or STOP BANG questionnaires.

The quantification of daytime sleepiness can potentially be of crucial importance both for diagnostic procedures and for the assessment of the use of therapeutic measures.

ELIGIBILITY:
Inclusion criteria for patients

* Age 18-80 years
* Written informed consent to participate in this study
* Patients with a clinical suspicion of sleep apnea

Exclusion criteria for patients:

* Age <18 years
* Lack of consent to participate in the study
* Lack of willingness and ability to participate in the study
* Pregnancy and breast feeding period

Inclusion criteria for healthy subjects:

* Age 18-45 years
* no internal or psychiatric illness requiring therapy
* not long-term drug therapy
* no known sleep apnea.
* Written consent to participate in this study

Exclusion criteria for healthy subjects:

* Patients with sleep apnea
* Age <18 years or ≥ 45 years
* Lack of consent to participate in the study
* Pregnancy and breast feeding period
* Lack of willingness and ability to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with the clinical suspicion of sleep apnea and healthy subject
  The healthy subjects will be recruited at the Lung and Allergy Centre, Practice for Internal Medicine, Pneumology, Allergology, Sleep and Sports Medicine Neuss in the clinical routine. The patients are from the Lung and Allergy Centre, Practice for Internal Medicine, Pneumology, Allergology, Sleep and Sports Medicine in Neuss and from the Div. of Cardiology, Pulmonary Disease and Vascular Medicine from the University Hospital Düsseldorf.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of Sleep Apnea | at Baseline
  the degree of daytime sleepiness can predict the presence of sleep apnea the degree of daytime sleepiness can predict the presence of sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof. Dr., Study Chair — Heinrich-Heine University, Duesseldorf
Locations (2):
- Germany (2):
  - Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia
  - Lung and Allergy Centre, Neuss, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided